CLINICAL TRIAL: NCT04593706
Title: Comparison of the Efficacy of Different Steroids in the Treatment of Abnormal Scars (Keloids, Hypertrophic Scars)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0542-19-TLV
Record Dates: First submitted 2020-07-29; First posted 2020-10-20 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-08

CONDITIONS: Keloid; Hypertrophic Scar; Scars; Scarring
MeSH Terms: conditions — Keloid; Cicatrix, Hypertrophic; Cicatrix | interventions — betamethasone acetate; betamethasone sodium phosphate; dexamethasone 21-phosphate; Methylprednisolone Acetate; Triamcinolone Acetonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- keloids (Active Comparator): each patient will be injection by all 4 steroids for comparison patients with 4 or more keloids will be injection with each steroid for different keloid
  Interventions: Drug: Betamethasone acetate + Betamethasone sodium phosphate; Drug: Dexamethasone sodium phosphate; Drug: Methylprednisolone acetate; Drug: Triamcinolone acetonide
- hypertrophic scars (Active Comparator): each patient will be injection by all 4 steroids for comparison patients with a 11 cm hypertrophic scar will be injected by all 4 steroids along the scar with a 1 cm distance between each steroid
  Interventions: Drug: Betamethasone acetate + Betamethasone sodium phosphate; Drug: Dexamethasone sodium phosphate; Drug: Methylprednisolone acetate; Drug: Triamcinolone acetonide

INTERVENTIONS:
Drug: Betamethasone acetate + Betamethasone sodium phosphate — the steroid will be injected to either a keloid or a 1.5 c"m of the 11 c"m hypertrophic scar
Drug: Dexamethasone sodium phosphate — the steroid will be injected to either a keloid or a 1.5 c"m of the 11 c"m hypertrophic scar
Drug: Methylprednisolone acetate — the steroid will be injected to either a keloid or a 1.5 c"m of the 11 c"m hypertrophic scar
Drug: Triamcinolone acetonide — the steroid will be injected to either a keloid or a 1.5 c"m of the 11 c"m hypertrophic scar

SUMMARY:
Comparison of the Efficacy of Different Steroids in the Treatment of Abnormal Scars (Keloids and hypertrophic Scars)

DETAILED DESCRIPTION:
On a yearly basis, millions develop different skin scarring. These scars are a public reminder of the traumatic incident, past or present disease or a surgery which caused them.

Scarring is a common consequence of wound healing process, and it is one of the most complex biological processes in human. This healing process is affected by numerous factors and thus can be disrupted, leading to pathological scarring.

Pathological scarring is common in people with genetic predisposition, those undergone complex and massive surgeries, burns or those wounded in unsanitary environments. Apart from being aesthetically unpleasant, scars are associated with functional and psychosocial morbidities.

Despite clinical, pathologic and pathogenic differences between keloids and hypertrophic scars, treatments are similar.

Scars have a negative external impact causing social distress and impaired self-image, and as a consequence, low satisfaction rates following surgical and cosmetic procedures.

The first line treatment is monthly intralesional corticosteroid injections with a response rate of 50-100% and recurrence of 50%.

There are a few steroids available and used for abnormal scars treatment, including Celestone chronodose (Betamethasone acetate + Betamethasone sodium phosphate), Dexamethasone sodium phosphate, Methylprednisolone acetate, Methylprednisolone sodium succinate, Methylprednisolone hemisuccinate, Triamcinolone acetonide.

Steroids are different by their hydrophilic properties, potency and half-life, although the half-life of intralesional injections is not known. Inspite of being widely used, there have never been a comparative study of the different steroid treatments.

ELIGIBILITY:
Inclusion Criteria:

* 20 participants with at least 4 keloids
* 20 participants with a hypertrophic scar of at least 11 cm length

Exclusion Criteria:

* current or planned pregnancy
* breastfeeding women
* participants suffering from diabetes mellitus or coagulation disorders
* infection at planned injection sites
* systemic treatment of corticosteroids, 5-fluorouracil
* known allergy to any of the following: Betamethasone acetate + Betamethasone sodium phosphate, Triamcinolone acetonide, Dexamethasone sodium phosphate, Methylprednisolone acetate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Patient and Observer Scar Assessment Scale (POSAS) | enrollment, data will be reported through study completion an average of 1 year
  For the Observer Scar Assessment Scale (OSAS), the investigators score the following parameters of each part of the scar on a scale ranging from 1 (normal skin) to 10 (worst scar imagin¬able): 'vascularization', 'pigmentation', 'thickness', 'relief', and 'pliability'. The total score on the OSAS is the sum of the scores of each item, yielding a total score ranging from 6 (best) to 60 (worst). For the patient scar assessment scale (PSAS), the participants used a scale of 1 to 10 to answer questions relating to pain, itching, color, stiffness, irregularity and thickness. The total score on the PSAS was the sum of the scores of each item, yielding a total score ranging from 6 (best) to 60 (worst)
Patient and Observer Scar Assessment Scale (POSAS) | 3 months post last treatment, data will be reported through study completion an average of 1 year
  For the Observer Scar Assessment Scale (OSAS), the investigators score the following parameters of each part of the scar on a scale ranging from 1 (normal skin) to 10 (worst scar imagin¬able): 'vascularization', 'pigmentation', 'thickness', 'relief', and 'pliability'. The total score on the OSAS is the sum of the scores of each item, yielding a total score ranging from 6 (best) to 60 (worst). For the patient scar assessment scale (PSAS), the participants used a scale of 1 to 10 to answer questions relating to pain, itching, color, stiffness, irregularity and thickness. The total score on the PSAS was the sum of the scores of each item, yielding a total score ranging from 6 (best) to 60 (worst)
Patient and Observer Scar Assessment Scale (POSAS) | 6 months post last treatment, data will be reported through study completion an average of 1 year
  For the Observer Scar Assessment Scale (OSAS), the investigators score the following parameters of each part of the scar on a scale ranging from 1 (normal skin) to 10 (worst scar imagin¬able): 'vascularization', 'pigmentation', 'thickness', 'relief', and 'pliability'. The total score on the OSAS is the sum of the scores of each item, yielding a total score ranging from 6 (best) to 60 (worst). For the patient scar assessment scale (PSAS), the participants used a scale of 1 to 10 to answer questions relating to pain, itching, color, stiffness, irregularity and thickness. The total score on the PSAS was the sum of the scores of each item, yielding a total score ranging from 6 (best) to 60 (worst)

SECONDARY OUTCOMES:
Visual analogue scale (pain scale) | at each of the three treatment appointments, data will be reported through study completion an average of 1 year
  1 - paineless, 10- extremely painfull
Dermatologist's assessment | 3 months post last treatment, data will be reported through study completion an average of 1 year
  0- no change, 1-minor change <5%, 2-Mild change - 25-50%, 3- Moderate Change 50-75%, 4-Significant change > 75%
3D camera | 3 months post last treatment, data will be reported through study completion an average of 1 year
  improvement percentage of scar volume
Participant's assessment | 3 months post last treatment, data will be reported through study completion an average of 1 year
  0- no change, 1-minor change <5%, 2-Mild change - 25-50%, 3- Moderate Change 50-75%, 4-Significant change > 75%
Dermatologist's assessment | 6 months post last treatment, data will be reported through study completion an average of 1 year
  0- no change, 1-minor change <5%, 2-Mild change - 25-50%, 3- Moderate Change 50-75%, 4-Significant change > 75%
3D camera | 6 months post last treatment, data will be reported through study completion an average of 1 year
  improvement percentage of scar volume
Participant's assessment | 6 months post last treatment, data will be reported through study completion an average of 1 year
  0- no change, 1-minor change <5%, 2-Mild change - 25-50%, 3- Moderate Change 50-75%, 4-Significant change > 75%